CLINICAL TRIAL: NCT06584734
Title: Effect of Intradialytic Exercise on Left Ventricular Diastolic Function in Hemodialysis Patients
Acronym: EXE-HDF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PT-23-1378
Record Dates: First submitted 2024-08-29; First posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Renal Dialysis; Hemodiafiltration; Diastolic Dysfunction; Kidney Failure; Resistance Training; Quality of Life
Keywords: Hemodiafiltration; Intradialytic Exercise; Diastolic Disfunction; Resistance Training
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Masking Description: There is no masking, patient is his own compared subject
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients in hemodiafiltration (Other): Patients having hemodiafiltration sessions 3 times a week, they used to do intradyalitic exercise but this exercise was neither measured, quantified, or supervised, so they were withdrawn from this exercise for three months and after this time, structured, measured and supervised intradialytic exercise was introduced.
  Interventions: Other: Not exercise; Other: Exercise during hemodiafiltration session

INTERVENTIONS:
Other: Not exercise — Patients were withdrawn from the exercise they had previously been doing during their hemodiafiltration sessions.
Other: Exercise during hemodiafiltration session — Exercise with cycle ergometers during hemodiafiltration session, intensity was measure with power meters in Watts units.

SUMMARY:
Introduction: Cardiovascular diseases are the leading cause of morbidity and mortality in hemodialysis patients, primarily due to structural cardiac changes that lead to diastolic dysfunction. Furthermore, this population has a high prevalence of sedentary behavior and increased mortality associated with it. Recent studies have implemented exercise regimens in the chronic kidney disease population, demonstrating improvements in various parameters related to cardiovascular disease.

Objectives: To evaluate the effect of implementing systematic intradialytic exercise on left ventricular diastolic function.

Materials and Methods: This is a quasi-experimental study (before-and-after type) that will be conducted in two phases. In the first phase (rest), both incident and prevalent hemodialysis patients will receive treatment for 3 months. A baseline echocardiogram will be performed and then repeated at the end of the first phase to determine left ventricular diastolic function parameters. The second phase of the study (intradialytic exercise) will take place during the following 3 months, with an echocardiogram performed at the beginning and end of this phase. Systematic, prescribed, and supervised intradialytic aerobic exercise (intradialytic pedaling) will be implemented. Additionally, a 6-minute walk test and a validated physical activity questionnaire will be administered monthly during both phases of the study.

DETAILED DESCRIPTION:
Left Ventricular Diastolic Function worsens during the hemodialysis session mainly due to preload effects. However, studies in patients with advanced CKD (pre-dialysis) have shown benefits in diastolic function when subjected to exercise programs. Based on this, implementing a standardized and protocolized exercise regimen during the hemodialysis session could provide cardiovascular benefits, specifically in terms of improving left ventricular diastolic function in this population.

The implementation of intradialytic exercise in the hemodialysis unit of our Institute began in 2004. However, there is no standardized or systematic process for intradialytic exercise.

This leads us to ask the following question: What is the effect of performing systematic intradialytic exercise on the echocardiographic parameters of left ventricular diastolic function in hemodialysis patients?

Methodology

Study Design:

* Non-randomized clinical trial (quasi-experimental, before-and-after study).
* Purpose: Analytical
* Temporal sequence: Longitudinal
* Control of study factor assignment: Experimental
* Chronology: Prospective

Study Population Description:

The target population is patients with chronic kidney disease who are currently in the unit and/or those who join the hemodialysis program at the National Institute of Cardiology (prevalent and incident hemodialysis patients).

Eligible Population:

Patients with chronic kidney disease, both prevalent and incident in hemodialysis, who are treated in the hemodialysis unit at the National Institute of Cardiology, with left ventricular diastolic function determined by echocardiographic measurement within a 6-month period from September 2023 to September 2024.

Once the inclusion criteria are met, a baseline transthoracic echocardiogram will be performed to determine and record the parameters that evaluate left ventricular diastolic function. If the patient presents any degree of diastolic dysfunction, the study will begin with a 3-month hemodialysis period without exercise. All echocardiograms will be performed before the first dialysis session of the week (Monday or Tuesday according to the patient's session schedule). At the end of the 3 months, a final transthoracic echocardiogram will be performed. The second phase of the study, which consists of hemodialysis with intradialytic exercise for 3 months, will then begin, and at the end of this period, another final transthoracic echocardiogram will be performed to determine diastolic function parameters. All echocardiograms will be performed before the first dialysis session of the week (Monday or Tuesday according to the patient's session schedule).

Evaluation of Intradialytic Exercise:

The prescription of intradialytic exercise will be based on the FITT-VP protocol, validated by the American College of Sports Medicine, which consists of the following points:

* F: Frequency
* I: Intensity
* T: Time
* T: Type
* V: Volume or amount of exercise
* P: Progression

Based on this, a cardiopulmonary exercise test will be conducted by a sports medicine expert for all patients. Based on the results and according to Skinner's three-phase model, the prescribed workload will be determined by the first ventilatory threshold (VT1), which lies between training zones 1 and 2. Adjustments will be made according to the FITT-VP points as follows:

Frequency:

* 2 times a week during the hemodialysis session (incident patients)
* 3 times a week during the hemodialysis session (prevalent patients)

Intensity: Low (no resistance), maintaining the VT1 watts throughout the session.

Time: Initially 45 minutes, increasing by 5 minutes each week, reaching 1 hour 30 minutes of exercise at the end of the study phase.

Type: Aerobic (stationary cycling).

Volume: Continuous pedaling during the hemodialysis session with work monitored in watts using power meters.

Progression: Progress will be recorded during the intradialytic exercise period.

Intradialytic exercise will be performed with a stationary bicycle model Urban fit PRO SH-612. Power meters (Favero Assioma UNO) will be inserted into the pedals and connected to a cycle computer (iGPSPORT BSC100S) to measure the workload in watts. The intradialytic exercise program will consist of pedaling during the hemodialysis session, with heart rate reserve monitored using the modified Karvonen method ((HRmax-HRrest)×(40-80%)+ HRrest) and Borg's Rating of Perceived Exertion Scale. A record will be kept for each session. Exercise prescription will be supervised by a sports medicine specialist, along with two medical interns trained in cardiopulmonary exercise testing, who will be responsible for registering and supervising the intradialytic exercise program.

Evaluation of Diastolic Function:

Diastolic function will be measured based on the international recommendations of the American and European Societies of Echocardiography published in 2016. The two-dimensional echocardiography study will be performed by two experienced cardiologists with current certification in echocardiography, using the Vivid Q GE ultrasound machine with a 3.5 MHz transducer. The following measurements will be taken:

* Early transmitral flow velocity (E wave)
* Late diastolic transmitral flow velocity (A wave)
* E/A ratio in an apical 4-chamber view with pulsed Doppler, placing the sample volume at the tips of the mitral valve leaflets.
* Tissue Doppler imaging (TDI) will be performed in an apical 4-chamber view to determine septal e' and lateral e' waves, with the pulsed Doppler sample volume placed 5 mm in the medial and lateral regions of the mitral annulus. The E/e' ratio will be calculated.
* Left atrial (LA) volume will be measured in an apical 4-chamber view and indexed to body surface area.
* Tricuspid regurgitation velocity (TR) will be measured with continuous Doppler in the apical 4-chamber approach focused on the right ventricle.

Based on these parameters, measurements will be categorized into grades of diastolic dysfunction (1, 2, 3, or indeterminate) according to current guidelines for patients with either reduced or preserved LVEF as appropriate. Left atrial strain will be measured using tissue Doppler in an apical 4-chamber view with the speckle tracking method.

6-Minute Walk Test: The test will be conducted on the first day of the hemodialysis session (Monday or Tuesday) before the session, every 4 weeks. The test will be performed based on the guidelines of the American and European Thoracic Societies by two medical interns trained to administer the test.

General Practice Physical Activity Questionnaire (GPPAQ):

The GPPAQ questionnaire will be administered to each patient at the beginning and every 4 weeks thereafter, on the same day and before the 6-minute walk test. The GPPAQ is a self-administered questionnaire for adults consisting of 3 questions. The first question measures the type and amount of physical activity (PA) at work, the second asks about the time spent on different types of PA during the last week, and the third asks about the usual walking pace. The scoring system classifies patients into 4 levels of PA: inactive (sedentary work and no physical exercise or cycling), moderately inactive (sedentary work and <1 hour of physical exercise or cycling, or standing work without physical exercise or cycling), moderately active (sedentary work and 1-2.9 hours/week of physical exercise or cycling, or standing work and <1 hour/week of physical exercise or cycling, or physically active work without physical exercise or cycling), and active (sedentary work and ≥3 hours/week of physical exercise or cycling, or standing work and 1-2.9 hours/week of physical exercise or cycling, or physically active work and <1 hour of physical exercise or cycling, or work with vigorous PA).

ELIGIBILITY:
Inclusion Criteria:

* Adults > 17 years
* Both genders
* Patients currently enrolled in the hemodialysis program at the National Institute of Cardiology unit
* Patients entering the hemodialysis program at the National Institute of Cardiology unit
* Patients with a good echocardiographic window that allows for the determination of parameters evaluating left ventricular diastolic function
* Patients capable of performing stationary cycling during hemodialysis sessions
* Patients who agree to participate in the study

Exclusion Criteria:

* Patients who have had a major cardiovascular event (MI, stroke) in the 3 months prior to the start of the study
* Patients who have visited the emergency room for symptoms of decompensated heart failure in the 3 months prior to the start of the study
* Patients diagnosed with atrial fibrillation and/or atrial flutter
* Patients with a mechanical mitral valve prosthesis
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-09-17 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of diastolic dysfunction | Basal measure (Previous exercise), 3 months after withdrawn of previous exercise during dialysis, 3 months after structured exercise during dialysis
  Diastolic function will be assessed following the 2016 guidelines from the American and European Societies of Echocardiography. The study will be performed by certified cardiologists using a Vivid Q GE ultrasound machine with a 3.5 MHz transducer. Key measurements include early (E wave) and late (A wave) transmitral flow velocities, E/A ratio, and tissue Doppler imaging (TDI) to determine septal and lateral e' waves. The E/e' ratio will be calculated. Left atrial (LA) volume will be measured and indexed to body surface area. Tricuspid regurgitation (TR) velocity will be assessed using continuous Doppler. Based on these parameters, diastolic dysfunction will be classified into grades 1, 2, 3, or indeterminate, according to current guidelines, considering whether the ejection fraction (EF) is reduced or preserved. The determination of left atrial strain will be performed using tissue Doppler imaging in an apical 4-chamber view with the speckle tracking method.

SECONDARY OUTCOMES:
6 minute walk test | Basal measure (Previous exercise), 3 months after withdrawn exercise, 3 months after structured exercise
  The test will be performed on the first day of the hemodialysis session (Monday or Tuesday) before the dialysis session, with a frequency of every 4 weeks. The test will be conducted based on the guidelines of the American and European Thoracic Societies by two medical interns, who are trained to perform the test
VO2 max | 3 months after withdrawn of previous exercise, 3 months after structures exercise
  Cardiopulmonary exercise test with cycle ergometer will be made by a specialized sports physician to the patients to asses training zones, in this test we will measure any improvement on VO2max (ml/min/kg)

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Cardiología Ignacio Chávez, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cusumano AM, Rosa-Diez GJ, Gonzalez-Bedat MC. Latin American Dialysis and Transplant Registry: Experience and contributions to end-stage renal disease epidemiology. World J Nephrol. 2016 Sep 6;5(5):389-97. doi: 10.5527/wjn.v5.i5.389. PMID 27648403
- [Background] Vasquez-Jimenez E, Madero M. Global Dialysis Perspective: Mexico. Kidney360. 2020 Apr 20;1(6):534-537. doi: 10.34067/KID.0000912020. eCollection 2020 Jun 25. No abstract available. PMID 35368596
- [Background] Mendez-Duran A, Ignorosa-Luna MH, Perez-Aguilar G, Rivera-Rodriguez FJ, Gonzalez-Izquierdo JJ, Davila-Torres J. [Current status of alternative therapies renal function at the Instituto Mexicano del Seguro Social]. Rev Med Inst Mex Seguro Soc. 2016 Sep-Oct;54(5):588-93. Spanish. PMID 27428340
- [Background] Collins AJ, Foley RN, Herzog C, Chavers B, Gilbertson D, Ishani A, Kasiske B, Liu J, Mau LW, McBean M, Murray A, St Peter W, Guo H, Gustafson S, Li Q, Li S, Li S, Peng Y, Qiu Y, Roberts T, Skeans M, Snyder J, Solid C, Wang C, Weinhandl E, Zaun D, Arko C, Chen SC, Dalleska F, Daniels F, Dunning S, Ebben J, Frazier E, Hanzlik C, Johnson R, Sheets D, Wang X, Forrest B, Constantini E, Everson S, Eggers P, Agodoa L. US Renal Data System 2010 Annual Data Report. Am J Kidney Dis. 2011 Jan;57(1 Suppl 1):A8, e1-526. doi: 10.1053/j.ajkd.2010.10.007. No abstract available. PMID 21184928
- [Background] Johansen KL, Chertow GM, Foley RN, Gilbertson DT, Herzog CA, Ishani A, Israni AK, Ku E, Kurella Tamura M, Li S, Li S, Liu J, Obrador GT, O'Hare AM, Peng Y, Powe NR, Roetker NS, St Peter WL, Abbott KC, Chan KE, Schulman IH, Snyder J, Solid C, Weinhandl ED, Winkelmayer WC, Wetmore JB. US Renal Data System 2020 Annual Data Report: Epidemiology of Kidney Disease in the United States. Am J Kidney Dis. 2021 Apr;77(4 Suppl 1):A7-A8. doi: 10.1053/j.ajkd.2021.01.002. No abstract available. PMID 33752804
- [Background] Di Lullo L, House A, Gorini A, Santoboni A, Russo D, Ronco C. Chronic kidney disease and cardiovascular complications. Heart Fail Rev. 2015 May;20(3):259-72. doi: 10.1007/s10741-014-9460-9. PMID 25344016
- [Background] Go AS, Chertow GM, Fan D, McCulloch CE, Hsu CY. Chronic kidney disease and the risks of death, cardiovascular events, and hospitalization. N Engl J Med. 2004 Sep 23;351(13):1296-305. doi: 10.1056/NEJMoa041031. PMID 15385656
- [Background] Levey AS, Eckardt KU, Tsukamoto Y, Levin A, Coresh J, Rossert J, De Zeeuw D, Hostetter TH, Lameire N, Eknoyan G. Definition and classification of chronic kidney disease: a position statement from Kidney Disease: Improving Global Outcomes (KDIGO). Kidney Int. 2005 Jun;67(6):2089-100. doi: 10.1111/j.1523-1755.2005.00365.x. PMID 15882252
- [Background] Gupta S, Dev V, Kumar MV, Dash SC. Left ventricular diastolic function in end-stage renal disease and the impact of hemodialysis. Am J Cardiol. 1993 Jun 15;71(16):1427-30. doi: 10.1016/0002-9149(93)90604-b. PMID 8517388
- [Background] Ruffmann K, Mandelbaum A, Bommer J, Schmidli M, Ritz E. Doppler echocardiographic findings in dialysis patients. Nephrol Dial Transplant. 1990;5(6):426-31. doi: 10.1093/ndt/5.6.426. PMID 2122318
- [Background] Antlanger M, Aschauer S, Kopecky C, Hecking M, Kovarik JJ, Werzowa J, Mascherbauer J, Genser B, Saemann MD, Bonderman D. Heart Failure with Preserved and Reduced Ejection Fraction in Hemodialysis Patients: Prevalence, Disease Prediction and Prognosis. Kidney Blood Press Res. 2017;42(1):165-176. doi: 10.1159/000473868. Epub 2017 Apr 11. PMID 28395286
- [Background] Sarafidis PA, Kamperidis V, Loutradis C, Tsilonis K, Mpoutsiouki F, Saratzis A, Giannakoulas G, Sianos G, Karvounis H. Haemodialysis acutely deteriorates left and right diastolic function and myocardial performance: an effect related to high ultrafiltration volumes? Nephrol Dial Transplant. 2017 Aug 1;32(8):1402-1409. doi: 10.1093/ndt/gfw345. PMID 27738230
- [Background] Drighil A, Madias JE, Mathewson JW, El Mosalami H, El Badaoui N, Ramdani B, Bennis A. Haemodialysis: effects of acute decrease in preload on tissue Doppler imaging indices of systolic and diastolic function of the left and right ventricles. Eur J Echocardiogr. 2008 Jul;9(4):530-5. doi: 10.1093/ejechocard/jen125. Epub 2008 Mar 27. PMID 18490307
- [Background] Nagueh SF, Smiseth OA, Appleton CP, Byrd BF 3rd, Dokainish H, Edvardsen T, Flachskampf FA, Gillebert TC, Klein AL, Lancellotti P, Marino P, Oh JK, Popescu BA, Waggoner AD. Recommendations for the Evaluation of Left Ventricular Diastolic Function by Echocardiography: An Update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. J Am Soc Echocardiogr. 2016 Apr;29(4):277-314. doi: 10.1016/j.echo.2016.01.011. No abstract available. PMID 27037982
- [Background] Malik J, Kudlicka J, Valerianova A, Kovarova L, Kmentova T, Lachmanova J. Diastolic dysfunction in asymptomatic hemodialysis patients in the light of the current echocardiographic guidelines. Int J Cardiovasc Imaging. 2019 Feb;35(2):313-317. doi: 10.1007/s10554-019-01564-2. Epub 2019 Feb 27. PMID 30815807
- [Background] Maufrais C, Josse M, Patrier L, Grandperrin A, Isnard M, Turc-Baron C, Nottin S, Mandigout S, Cristol JP, Obert P. Cardioprotective effect of intradialytic exercise on left atrial mechanics. Am J Physiol Renal Physiol. 2024 May 1;326(5):F694-F703. doi: 10.1152/ajprenal.00380.2023. Epub 2024 Mar 21. PMID 38511221
- [Background] Baker LA, March DS, Wilkinson TJ, Billany RE, Bishop NC, Castle EM, Chilcot J, Davies MD, Graham-Brown MPM, Greenwood SA, Junglee NA, Kanavaki AM, Lightfoot CJ, Macdonald JH, Rossetti GMK, Smith AC, Burton JO. Clinical practice guideline exercise and lifestyle in chronic kidney disease. BMC Nephrol. 2022 Feb 22;23(1):75. doi: 10.1186/s12882-021-02618-1. No abstract available. PMID 35193515
- [Background] Greenwood SA, Lindup H, Taylor K, Koufaki P, Rush R, Macdougall IC, Mercer TH. Evaluation of a pragmatic exercise rehabilitation programme in chronic kidney disease. Nephrol Dial Transplant. 2012 Oct;27 Suppl 3:iii126-34. doi: 10.1093/ndt/gfs272. Epub 2012 Jul 10. PMID 22785111
- [Background] Beddhu S, Baird BC, Zitterkoph J, Neilson J, Greene T. Physical activity and mortality in chronic kidney disease (NHANES III). Clin J Am Soc Nephrol. 2009 Dec;4(12):1901-6. doi: 10.2215/CJN.01970309. Epub 2009 Oct 9. PMID 19820134
- [Background] Wilkinson TJ, Clarke AL, Nixon DGD, Hull KL, Song Y, Burton JO, Yates T, Smith AC. Prevalence and correlates of physical activity across kidney disease stages: an observational multicentre study. Nephrol Dial Transplant. 2021 Mar 29;36(4):641-649. doi: 10.1093/ndt/gfz235. PMID 31725147
- [Background] Oh W, Cho M, Jung SW, Moon JY, Lee SH, Hwang YC, Kim YG. High physical activity alleviates the adverse effect of higher sedentary time on the incidence of chronic kidney disease. J Cachexia Sarcopenia Muscle. 2023 Feb;14(1):622-631. doi: 10.1002/jcsm.13167. Epub 2022 Dec 25. PMID 36567072
- [Background] Pearson MJ, Mungovan SF, Smart NA. Effect of exercise on diastolic function in heart failure patients: a systematic review and meta-analysis. Heart Fail Rev. 2017 Mar;22(2):229-242. doi: 10.1007/s10741-017-9600-0. PMID 28229273
- [Background] Young HML, March DS, Graham-Brown MPM, Jones AW, Curtis F, Grantham CS, Churchward DR, Highton P, Smith AC, Singh SJ, Bridle C, Burton JO. Effects of intradialytic cycling exercise on exercise capacity, quality of life, physical function and cardiovascular measures in adult haemodialysis patients: a systematic review and meta-analysis. Nephrol Dial Transplant. 2018 Aug 1;33(8):1436-1445. doi: 10.1093/ndt/gfy045. PMID 29608708
- [Background] Graham-Brown MPM, March DS, Young R, Highton PJ, Young HML, Churchward DR, Dungey M, Stensel DJ, Bishop NC, Brunskill NJ, Smith AC, McCann GP, McConnachie A, Burton JO. A randomized controlled trial to investigate the effects of intra-dialytic cycling on left ventricular mass. Kidney Int. 2021 Jun;99(6):1478-1486. doi: 10.1016/j.kint.2021.02.027. Epub 2021 Apr 8. PMID 34023029
- [Background] Momeni A, Nematolahi A, Nasr M. Effect of intradialytic exercise on echocardiographic findings in hemodialysis patients. Iran J Kidney Dis. 2014 May;8(3):207-11. PMID 24878943
- [Background] Jeong JH, Biruete A, Fernhall B, Wilund KR. Effects of acute intradialytic exercise on cardiovascular responses in hemodialysis patients. Hemodial Int. 2018 Oct;22(4):524-533. doi: 10.1111/hdi.12664. Epub 2018 May 9. PMID 29745006
- [Background] Penny JD, Salerno FR, Brar R, Garcia E, Rossum K, McIntyre CW, Bohm CJ. Intradialytic exercise preconditioning: an exploratory study on the effect on myocardial stunning. Nephrol Dial Transplant. 2019 Nov 1;34(11):1917-1923. doi: 10.1093/ndt/gfy376. PMID 30590580
- [Background] Skinner JS, McLellan TM. The transition from aerobic to anaerobic metabolism. Res Q Exerc Sport. 1980 Mar;51(1):234-48. doi: 10.1080/02701367.1980.10609285. No abstract available. PMID 7394286
- [Background] Lucia A, Sanchez O, Carvajal A, Chicharro JL. Analysis of the aerobic-anaerobic transition in elite cyclists during incremental exercise with the use of electromyography. Br J Sports Med. 1999 Jun;33(3):178-85. doi: 10.1136/bjsm.33.3.178. PMID 10378070
- [Background] Karvonen J, Vuorimaa T. Heart rate and exercise intensity during sports activities. Practical application. Sports Med. 1988 May;5(5):303-11. doi: 10.2165/00007256-198805050-00002. PMID 3387734
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Nagueh SF, Khan SU. Left Atrial Strain for Assessment of Left Ventricular Diastolic Function: Focus on Populations With Normal LVEF. JACC Cardiovasc Imaging. 2023 May;16(5):691-707. doi: 10.1016/j.jcmg.2022.10.011. Epub 2023 Jan 11. PMID 36752445
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180